CLINICAL TRIAL: NCT01923103
Title: Natural Disease Progress of Dupuytren Disease
Acronym: DD
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, D.C. Broekstra, PhD, University Medical Center Groningen
Other Study IDs: NDPDD
Record Dates: First submitted 2013-08-09; First posted 2013-08-14 (Estimated); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Dupuytren Contracture; Disease Progression
MeSH Terms: conditions — Dupuytren Contracture; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No

SUMMARY:
Dupuytren disease (DD) is a progressive fibromatosis of the palmar fascias of the hand and fingers, which may lead to extension deficits of the fingers. The disease can be very disabling in moderate and severe cases, whereby performing normal daily activities can become very problematic. The aetiology and pathogenesis are not completely understood. There is a genetic disposition and it is influenced by environmental factors. The disease is especially prevalent in white males of Northern European descent above 50 years of age. There is paucity of knowledge about the natural progression of the disease. Several studies have been conducted on progression of disease and from these studies it becomes obvious that the disease is progressive over several years. However, in most studies only one moment of follow-up has taken place, so the course of the progression over time is unknown.

The aim of this study is to enhance our knowledge on the natural disease progression of DD at different stages.

DETAILED DESCRIPTION:
Objective:

* Primary objective: To study natural disease progress of Dupuytren Disease (DD) in different stages of disease in males and females above 18 years of age.
* Secondary objectives:

  1. To study the effect of potential risk factors for DD on natural disease progress.
  2. To study at what stage of disease patients with DD experience problems in daily life.
  3. To study the incidence and course of recurrent disease. Primary Hypothesis: The natural course of disease is an exponential function of time.
  4. To study the intrarater reliability of the measurements

  f. To determine whether the echogenicity of the nodules can predict progression g. To determine whether extension deficit measurements can be replaced by measurements of extension, and whether this will facilitate the statistical analysis h. To determine the association between passive and active measurements of extension and extension deficit, and to see whether active measurements can be derived from passive measurements and vice versa.
* Study design: The study is designed as a prospective observational pilot study with a follow-up of 10 years.
* Study population: Males and females above 18 years of age with all stages of primary Dupuytren's disease in at least one hand
* Main study parameters/endpoints: The natural course of progression of DD measured as the increase or decrease in size of nodules and cords in millimetres and/or increase of total passive extension deficit in degrees, from baseline to endpoint.
* Secondary study parameters:

  1. Patient-reported hand function (Michigan Hand Outcomes Questionnaire (MHOQ), Patient-Rated Wrist/Hand Evaluation (PRWHE) and Unité Rhumatologique des Affections de la Main (URAM) scale
  2. incidence and course of recurrent disease
  3. disease activity (ultrasonography and tonometry)
* Procedure Patients visit the outpatient clinic every 6 months (first 5 years of follow-up) and later on every 12 months (last 5 years of follow-up) for an anamnestic interview, physical examination of the hands, ultrasonography, tonometry and for filling out the PROMs.

ELIGIBILITY:
Inclusion Criteria:

* Patients (> 18 years of age) with primary Dupuytren's disease in all Tubiana stages
* Operated hands of patients with primary Dupuytren's disease on the contra lateral hand

Exclusion Criteria:

* Patients who are incapable of giving consent
* Patients who are not able or not willing to visit the UMCG for follow-up
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Dupuytren Disease who participated in prior studies and patients from the outpatient clinic
Sampling Method: Non-Probability Sample
Enrollment: 261 (Actual)
Dates: Start 2012-06-22 (Actual); Primary Completion 2023-03 (Actual); Study Completion 2023-03-20 (Actual)

PRIMARY OUTCOMES:
The course of DD: passive and active extension deficit and dimension of palpable nodules and cords | every 6-12 months
  Active and passive extension deficit is measured with a goniometer at joint level Dimension of nodules and cords is measured using a tumorimeter

SECONDARY OUTCOMES:
Disease activity: Echogenicity and nodule hardness | every 12 months, starting from 2016 (ultrasound) and 2018 (tonometry)
  Activity of a nodule is determined by 1) echogenicity of the ultrasound image in sagittal and transversal plane, 2) hardness of the nodule determined by tonometry
Patient-reported hand function: MHQ, PRWHE and URAM | every 6-12 months
  To study what problems patients with DD experience in daily life, PROMs are used. MHQ and PRWHE in the first 2 years, URAM later on

CONTACTS AND LOCATIONS:
Overall Officials: Paul MN Werker, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No
There is no plan available, but we are open for collaboration